CLINICAL TRIAL: NCT00529126
Title: A Phase 2 Multicenter, Randomized, Double-blind, Parallel-group, Active-control, Dose-ranging Study to Evaluate the Safety and Efficacy of a Single Administration of SKY0402 for Prolonged Postoperative Analgesia in Subject Undergoing Hemorrhoidectomy
Brief Title: Phase 2 Dose-Ranging Study of SKY0402 for Prolonged Postoperative Analgesia in Subject Undergoing Hemorrhoidectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SKY0402C209
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Results first posted 2013-08-06 (Estimated); Last update posted 2021-03-04 (Actual); Status verified 2021-02

CONDITIONS: Postoperative Pain
Keywords: hemorrhoidectomy; pain; Postoperative; analgesia
MeSH Terms: conditions — Pain, Postoperative; Pain; Agnosia | interventions — Bupivacaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- SKY0402 high dose (Experimental): SKY0402, single administration
  Interventions: Drug: SKY0402
- SKY0402 middle dose (Experimental): SKY0402, single administration
  Interventions: Drug: SKY0402
- SKY0402 low dose (Experimental): SKY0402, single administration
  Interventions: Drug: SKY0402
- Bupivacaine HCl (Active Comparator): Bupivacaine HCl
  Interventions: Drug: Bupivacaine HCl

INTERVENTIONS:
Drug: SKY0402 — SKY0402
  Other Names: EXPAREL
  Arms: SKY0402 high dose; SKY0402 low dose; SKY0402 middle dose
Drug: Bupivacaine HCl — Bupivacaine HCl
  Other Names: Marcaine 0.25% with epinephrine 1:200,000
  Arms: Bupivacaine HCl

SUMMARY:
Phase 2 study to evaluate three dose levels of SKY0402 compared with 75 mg of bupivacaine HCl.

DETAILED DESCRIPTION:
Effective postoperative pain control is a critical element in patient recovery, as the majority of patients may experience significant pain, particularly in the first few days following surgery. Appropriate postoperative pain management contributes to improved healing, faster patient mobilization, shortened hospital stays, and reduced healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years of age and older at the Screening Visit.
2. Applies to female subjects only: Postmenopausal, surgically sterile, or willing to use acceptable means of contraception for at least 30 days after surgery including any of the following: hormonal contraceptives (e.g., oral, injectable, implantable starting at least 30 days before study drug administration), effective double-barrier methods (e.g., condoms with spermicide), intrauterine device, lifestyle with a personal choice of abstinence, nonheterosexual lifestyle, or a strictly monogamous relationship with a partner who has had a vasectomy.
3. Scheduled to undergo 2- or 3-column excisional hemorrhoidectomy under general anesthesia using Milligan Morgan or Ferguson-type techniques, including modified approaches with specialized instruments, such as LigaSure™ or harmonic scalpel, with a cumulative incision length of a minimum 3 cm.
4. American Society of Anesthesiology (ASA) Physical Class 1-3.
5. Able and willing to comply with all study visits and procedures.
6. Able to speak, read, and understand the language of the Informed Consent Form (ICF), study questionnaires, and other instruments used for collecting subject-reported outcomes, in order to enable accurate and appropriate responses to pain scales and other required study assessments.
7. Willing and capable of providing written informed consent.

Exclusion Criteria:

1. Pregnancy, nursing, or planning to become pregnant during the study or within one month after study drug administration.
2. Use of any of the following medications within the times specified before surgery:

   * Long-acting opioid medication within 3 days.
   * Any opioid medication within 24 hours.
3. Concurrent painful physical condition that may require analgesic treatment in the postoperative period for pain that is not surgically related and may confound the postoperative assessments (e.g., rheumatoid arthritis, chronic neuropathic pain).
4. Single-column hemorrhoidectomy or hemorrhoidectomy without an internal component.
5. Body weight less than 50 kilograms (110 pounds).
6. History of hypersensitivity or idiosyncratic reactions to amide-type local anesthetics or to opioid medication.
7. Contraindication to epinephrine, such as concurrent administration of monoamine oxidase (MAO) inhibitors or antidepressants of amitriptyline or imipramine types, conditions where the production or exacerbation of tachycardia could prove fatal (e.g., poorly controlled thyrotoxicosis or severe heart disease), or any other pathological conditions that might be aggravated by the effects of epinephrine.
8. Contraindications to any of the pain-control agents planned for postoperative use (e.g., acetaminophen [paracetamol], oxycodone, morphine, ketorolac).
9. Administration of an investigational drug within 30 days or 5 elimination half-lives of such investigational drug, whichever is longer, prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study.
10. History of, suspected, or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years.
11. Uncontrolled anxiety, schizophrenia, or other psychiatric disorder that, in the opinion of the Investigator, may interfere with study assessments or compliance.
12. Significant medical conditions or laboratory results that, in the opinion of the Investigator, indicate an increased vulnerability to study drugs and procedures, and expose the subject to an unreasonable risk as a result of participating in this clinical trial, such as: debilitating diseases, acute illnesses, hypotension, partial or complete conduction block, impaired cardiac function, untreated hypertension, advanced arteriosclerotic heart disease, cerebral vascular insufficiency, pre-existing abnormal neurological or neuromuscular disease (e.g., epilepsy, myasthenia gravis), advanced liver disease, severe renal impairment, advanced diabetes, comorbid conditions associated with an immunocompromised status, such as blood dyscrasias, HIV/AIDS, or recent chemotherapy.

    In addition, the subject will be ineligible to receive study drug if he or she meets the following criteria during surgery:
13. Any clinically significant event or condition uncovered during the surgery (e.g., excessive bleeding, acute sepsis) that might render the subject medically unstable or complicate the subject's postoperative course.
14. A cumulative incision length less than 3 cm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-09; Primary Completion 2007-12 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erol Onel, MD, Study Director — Pacira Pharmaceuticals, Inc
Locations (7):
- United States (4):
  - Accurate Clinical Trials, Inc., San Clemente, California
  - University of Miami/Jackson Memorial, Miami, Florida
  - The Women's Hospital of Texas, Houston, Texas
  - Multicare Health Systems Laboratories, Tacoma, Washington
- Georgia (3):
  - JSC Imereti Regional Clinical Hospital of the Name A. Dzotsenidze, Kutaisi
  - JSC K. Eristavi National Center of Experimental and Clinical Surgery, Tbilisi
  - Socieety with limited responsibility Proctology Center, Tbilisi

REFERENCES:
- [Derived] Dasta J, Ramamoorthy S, Patou G, Sinatra R. Bupivacaine liposome injectable suspension compared with bupivacaine HCl for the reduction of opioid burden in the postsurgical setting. Curr Med Res Opin. 2012 Oct;28(10):1609-15. doi: 10.1185/03007995.2012.721760. Epub 2012 Sep 3. PMID 22900785

RESULTS

PARTICIPANT FLOW:
Groups:
- SKY0402 High Dose (300mg): SKY0402 300mg single dose administered intraoperatively via local infiltration.
- SKY0402 Middle Dose (225mg): A single dose 225mg SKY0402 administered intraoperatively via local infiltration.
- SKY0402 Low Dose (75mg): A single dose 75mg SKY0402 administered intraoperatively via local infiltration.
- Bupivacaine HCl 75mg: A single dose of 75 mg bupivacaine administered intraoperatively via local infiltration
Period: Overall Study
Arm/Group | SKY0402 High Dose (300mg) | SKY0402 Middle Dose (225mg) | SKY0402 Low Dose (75mg) | Bupivacaine HCl 75mg
Started | 25 | 25 | 24 | 26
Completed | 25 | 25 | 24 | 26
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- SKY0402 High Dose; SKY0402 Middle Dose; SKY0402 Low Dose: A single dose of study drug was to be administered intraoperatively via local infiltration.
- Bupivacaine HCl: A single dose of 75 mg bupivacaine was to be administered intraoperatively via local infiltration
- Total: Total of all reporting groups
Arm/Group | SKY0402 High Dose | SKY0402 Middle Dose | SKY0402 Low Dose | Bupivacaine HCl | Total
Number analyzed (Participants) | 25 | 25 | 24 | 26 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 24 | 23 | 25 | 95
  >=65 years | 2 | 1 | 1 | 1 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (11.3) | 41.7 (11.2) | 42.2 (11.5) | 44.2 (10.6) | 43.4 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 9 | 7 | 11 | 30
  Male | 22 | 16 | 17 | 15 | 70
Region of Enrollment [Number; unit: participants]
  United States | 5 | 9 | 9 | 14 | 37
  Georgia | 20 | 16 | 15 | 12 | 63

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) of the Numeric Rating Scale (NRS) at Rest (NRS-R) Pain Intensity Scores From 0 Through 72 Hours
Description: To assess pain intensity at rest (NRS-R), the subject was to assume a resting position that did not exacerbate his or her postoperative pain. The subject was to rest in this position for at least 5 minutes before responding to the following question: "On a scale of 0 to 10, where 0=no pain and 10=worst possible pain, how much pain are you having right now?"
Time Frame: 0 to 72 hours
Measure: Mean (Standard Deviation); unit: units on a scale*hrs
Groups:
- SKY0402 300mg: A single dose of SKY0402 300mg administered intraoperatively via local infiltration.
- SKY0402 225mg: A single dose of SKY0402 225mg administered intraoperatively via local infiltration.
- SKY0402 75mg: A single dose of SKY0402 75mg administered intraoperatively via local infiltration.
Arm/Group | SKY0402 300mg | SKY0402 225mg | SKY0402 75mg | Bupivacaine HCl
Number analyzed (Participants) | 25 | 25 | 24 | 26
units on a scale*hrs | 175 (173) | 172 (146) | 225 (185) | 331 (175)

2. Secondary Outcome: Participants With Adverse Events Through 72 Hours or Serious Adverse Events Through 30 Days
Time Frame: Up to 30 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | SKY0402 High Dose | SKY0402 Middle Dose | SKY0402 Low Dose | Bupivacaine HCl
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 1/24 | 0/26
Other Adverse Events (participants affected / at risk) | 0/25 | 7/25 | 7/24 | 10/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SKY0402 High Dose (N=25) | SKY0402 Middle Dose (N=25) | SKY0402 Low Dose (N=24) | Bupivacaine HCl (N=26)
Rectal hemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SKY0402 High Dose (N=25) | SKY0402 Middle Dose (N=25) | SKY0402 Low Dose (N=24) | Bupivacaine HCl (N=26)
Constipation (Gastrointestinal disorders) | 0 (0) | 5 | 3 | 4
Nausea (Gastrointestinal disorders) | 0 (0) | 4 | 3 | 3
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No